CLINICAL TRIAL: NCT00906360
Title: A Phase I Trial of Concurrent Chemoradiation/Chemoreirradiation With Cetuximab (ERBITUX®), Sunitinib, and Accelerated Radiation in Patients With Locally Advanced/High-risk/Recurrent Poor Prognosis Head and Neck Cancer
Brief Title: Sunitinib, Cetuximab, and Radiation Therapy in Treating Patients With Locally Advanced or Recurrent Squamous Cell Carcinoma of the Head and Neck
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00279; UCIRB 16051B; CDR0000601544; UCIRB-16051B; N01CM62201 (NIH)
Record Dates: First submitted 2009-05-20; First posted 2009-05-21 (Estimated); Last update posted 2013-07-02 (Estimated); Status verified 2013-07

CONDITIONS: Metastatic Squamous Neck Cancer With Occult Primary Squamous Cell Carcinoma; Recurrent Metastatic Squamous Neck Cancer With Occult Primary; Recurrent Salivary Gland Cancer; Recurrent Squamous Cell Carcinoma of the Hypopharynx; Recurrent Squamous Cell Carcinoma of the Larynx; Recurrent Squamous Cell Carcinoma of the Lip and Oral Cavity; Recurrent Squamous Cell Carcinoma of the Nasopharynx; Recurrent Squamous Cell Carcinoma of the Oropharynx; Recurrent Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Recurrent Verrucous Carcinoma of the Larynx; Recurrent Verrucous Carcinoma of the Oral Cavity; Salivary Gland Squamous Cell Carcinoma; Stage III Salivary Gland Cancer; Stage III Squamous Cell Carcinoma of the Hypopharynx; Stage III Squamous Cell Carcinoma of the Larynx; Stage III Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage III Squamous Cell Carcinoma of the Nasopharynx; Stage III Squamous Cell Carcinoma of the Oropharynx; Stage III Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Stage III Verrucous Carcinoma of the Larynx; Stage III Verrucous Carcinoma of the Oral Cavity; Stage IV Salivary Gland Cancer; Stage IV Squamous Cell Carcinoma of the Hypopharynx; Stage IV Squamous Cell Carcinoma of the Larynx; Stage IV Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IV Squamous Cell Carcinoma of the Nasopharynx; Stage IV Squamous Cell Carcinoma of the Oropharynx; Stage IV Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Stage IV Verrucous Carcinoma of the Larynx; Stage IV Verrucous Carcinoma of the Oral Cavity; Tongue Cancer; Untreated Metastatic Squamous Neck Cancer With Occult Primary
MeSH Terms: conditions — Salivary Gland Neoplasms; Squamous Cell Carcinoma of Head and Neck; Tongue Neoplasms | interventions — Sunitinib; Radiotherapy, Conformal; Cetuximab

ARMS (1):
- Treatment (enzyme inhibitor and monoclonal antibody therapy) (Experimental): Patients receive sunitinib malate orally or by percutaneous gastrostomy tube once daily, cetuximab IV over 60-120 minutes once weekly, and undergo concurrent radiotherapy once or twice daily, 5 days a week, for 7-9 weeks in the absence of disease progression or unacceptable toxicity. Patients with persistent disease undergo surgical resection.
  Interventions: Drug: sunitinib malate; Other: pharmacological study; Radiation: 3-dimensional conformal radiation therapy; Biological: cetuximab

INTERVENTIONS:
Drug: sunitinib malate — Given orally or by percutaneous gastrostomy tube
  Other Names: SU11248; sunitinib; Sutent
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Radiation: 3-dimensional conformal radiation therapy — Undergo radiotherapy
  Other Names: 3D conformal radiation therapy; 3D-CRT
Biological: cetuximab — Given IV
  Other Names: C225; C225 monoclonal antibody; IMC-C225; MOAB C225; monoclonal antibody C225

SUMMARY:
This phase I trial is studying the side effects and best dose of sunitinib when given together with cetuximab and radiation therapy in treating patients with locally advanced or recurrent squamous cell carcinoma of the head and neck. Sunitinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving sunitinib together with cetuximab and radiation therapy may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety, the maximum tolerated dose, and the dose limiting toxicity of sunitinib malate when administered in combination with cetuximab and radiotherapy in patients with locally advanced, recurrent, or second primary poor prognosis, high-risk squamous cell carcinoma of the head and neck.

SECONDARY OBJECTIVES:

I. To describe the toxicity profile of this regimen. II. To explore the tolerability and feasibility of sunitinib malate when administered in combination with cetuximab and radiotherapy in these patients.

III. To assess the best overall response rate (complete and partial response) after completion of treatment.

IV. To assess the locoregional control rate. V. To assess the distant control rate. VI. To assess the pharmacokinetics of sunitinib malate delivered by percutaneous gastrostomy tube.

OUTLINE: This is a dose-escalation study of sunitinib malate.

Patients receive sunitinib malate orally or by percutaneous gastrostomy tube once daily, cetuximab IV over 60-120 minutes once weekly, and undergo concurrent radiotherapy once or twice daily, 5 days a week, for 7-9 weeks in the absence of disease progression or unacceptable toxicity. Patients with persistent disease undergo surgical resection.

*NOTE: *Patients may have resection prior to enrollment on protocol provided they have high-risk features for recurrence.

Some patients undergo blood sample collection at baseline and periodically during study for pharmacokinetic analysis of sunitinib malate and metabolites.

After completion of study treatment, patients are followed up periodically for up to 6 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed squamous cell carcinoma of the head and neck, meeting any of the following criteria:

  * Recurrent disease
  * Second primary locoregional recurrence* with no clinically measurable distant disease
  * Poor prognosis non-metastatic head and neck carcinoma (M0)
* Must have undergone radiotherapy as a component of prior treatment
* Not a candidate for surgical resection with curative intent

  * Patients with high-risk features at resection or following resection for recurrence are eligible
* Must have locoregional tumor amenable to radiotherapy or reirradiation with curative intent

  * Entire gross tumor recurrence volume must be able to be treated without exceeding a cumulative spinal cord dose of 50 Gy
* Unresected tumors must be measurable according to RECIST
* No known brain metastases
* ECOG performance status (PS) 0-2 OR Karnofsky PS 60-100%
* Life expectancy > 12 weeks
* WBC ≥ 3,000/mm^³
* ANC > 1,500/mm³
* Platelet count > 100,000/mm³
* Total bilirubin < 1.5 times upper limit of normal (ULN)
* INR and PTT ratio < 1.5
* AST and ALT ≤ 2.5 times ULN
* Creatinine normal OR creatinine clearance > 60 mL/min
* Urine protein no more than trace
* Hematocrit ≥ 28%
* Hemoglobin ≥ 9 g/dL
* QTc < 500 msec
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* The following patients are eligible provided they have New York Heart Association class II cardiac function on baseline ECHO and MUGA:

  * Asymptomatic on treatment
  * Prior anthracycline exposure
  * Prior central thoracic radiotherapy included the heart in the radiotherapy port
* No clinical evidence of active infection of any type, including hepatitis B or C virus

  * Infections controlled with therapy are allowed
  * Patients with hepatitis B or C on antiviral therapy with no detectable virus are allowed
* No immune deficiency and/or HIV positivity
* No history of allergic reactions attributed to compounds of similar chemical or biological composition to sunitinib malate
* No gastrointestinal tract disease or condition, including any of the following, that impairs ability to retain sunitinib tablets:

  * Inability to take oral medication or a requirement for IV alimentation
  * Prior surgical procedures affecting absorption
  * Active peptic ulcer disease
* None of the following conditions allowed:

  * Serious or nonhealing wound, ulcer, or bone fracture
  * Abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 28 days
* No significant concurrent medical or psychiatric illness which, in the opinion of the investigator, would interfere with the patient's ability to participate in the trial
* No active carotid artery involvement
* No history of documented thrombosis (pulmonary embolism within the past 12 months or deep vein thrombosis [DVT] within the past 6 months), known coagulopathies or thrombophilia, or evidence of DVT/thromboembolic event
* No history of the following cardiovascular conditions :

  * Myocardial infarction within the past 12 months
  * Cardiac arrhythmia or serious ventricular arrhythmia (ventricular fibrillation or ventricular tachycardia ≥ 3 beats in a row) within the past 12 months
  * Stable/unstable angina within the past 12 months
  * Symptomatic congestive heart failure within the past 12 months
  * Coronary/peripheral artery bypass graft or stenting within the past 12 months
  * No cerebral vascular disease, cerebrovascular accident (stroke), or transient ischemic attack within the past 6 months
  * QTc prolongation (QTc interval ≥ 500 msec)
  * New York Heart Association class III-IV congestive heart failure
  * Poorly controlled hypertension (i.e., systolic blood pressure [BP] ≥ 140 mm Hg or diastolic BP ≥ 90 mm Hg)
  * Other significant ECG abnormalities
* See Disease Characteristics
* Recovered from all prior radiotherapy and chemotherapy
* More than 4 months since prior radiotherapy to the head and neck
* More than 2 weeks since prior hormone replacement therapy or hormonal contraceptives
* More than 4 weeks since prior and no other concurrent investigational agents
* At least 1 month since prior surgery (unless ambulatory within 48 hours)
* At least 7 days since prior and no concurrent CYP3A4 inhibitors, including any of the following:

  * Azole antifungals (ketoconazole, itraconazole)
  * Clarithromycin
  * Erythromycin
  * Diltiazem
  * Verapamil
  * HIV protease inhibitors (indinavir, saquinavir, ritonavir, atazanavir, nelfinavir)
  * Delavirdine
* At least 12 days since prior and no concurrent CYP3A4 inducers, including any of the following:

  * Rifampin
  * Rifabutin
  * Carbamazepine
  * Phenobarbital
  * Phenytoin
  * St. John wort
  * Efavirenz
  * Tipranavir
* Concurrent coumarin-derivative anticoagulants (e.g., warfarin up to 2 mg daily) allowed for prophylaxis of thrombosis
* Concurrent use of medications known to affect the conductive system (e.g., beta-blockers, calcium channel blockers, or digoxin) allowed under investigator supervision
* No concurrent agent with proarrhythmic potential, including any of the following:

  * Terfenadine
  * Quinidine
  * Procainamide
  * Disopyramide
  * Sotalol
  * Probucol
  * Bepridil
  * Haloperidol
  * Risperidone
  * Indapamide
  * Flecainide
* No concurrent chronic steroid treatment for > 6 months (i.e., prednisolone doses > 10 mg/day or equivalent)
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No concurrent amifostine
* No concurrent commercial agent or therapy intended to treat head and neck cancer
* No other concurrent anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2008-07; Primary Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Maximum-tolerated dose (MTD) of sunitinib malate | Up to 7-9 weeks
  MTD is defined as the dose level immediately below the non-tolerated dose. The study will utilize a standard "3+3" design to determine the MTD. Dose limiting toxicities (DLTs) used for determining escalation of dose will be those occurring within the period of radiotherapy. Toxicity will be summarized by type and severity using the National Cancer Institute (NCI) Common Terminology Criteria.

SECONDARY OUTCOMES:
Objective tumor response rates | From the start of the treatment to up to 6 years
  Response will be evaluated in this study using the new international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) Committee. The efficacy analysis population (an exploratory analysis of those patients on study for the MTD) will consist of all subjects who received at least 1 dose of sunitinib. Ninety percent confidence intervals using the exact binomial distribution will be presented. Kaplan-Meier product limit curves will be calculated.
Locoregional control rates | Up to 6 years
  Ninety percent confidence intervals using the exact binomial distribution will be presented. Kaplan-Meier product limit curves will be calculated.
Disease control rates | Up to 6 years
  Ninety percent confidence intervals using the exact binomial distribution will be presented. Kaplan-Meier product limit curves will be calculated.
Locoregional recurrence rates | At 3 years
  Ninety percent confidence intervals using the exact binomial distribution will be presented. Kaplan-Meier product limit curves will be calculated.
Time to progression | From the date of registration to the date of progressive disease or death from any cause
  Time to progression using Kaplan-Meier product limit curves will be calculated.
Overall survival time | From the date of registration to the date of death or date of last patient contact if censored
  Overall survival using Kaplan-Meier product limit curves will be calculated.
Pharmacokinetics of sunitinib malate delivered by percutaneous gastrostomy tube | Prior to and up to 24 hours after the start of sunitinib malate

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Villaflor, Principal Investigator — University of Chicago Comprehensive Cancer Center
Locations (12):
- United States (12):
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Evanston CCOP-NorthShore University HealthSystem, Evanston, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Fort Wayne Medical Oncology and Hematology Inc - State Boulevard, Fort Wayne, Indiana
  - University of Maryland Greenebaum Cancer Center, Baltimore, Maryland
  - University of Michigan University Hospital, Ann Arbor, Michigan
  - Saint John's Mercy Medical Center, St Louis, Missouri
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin